CLINICAL TRIAL: NCT03465891
Title: Two-Arm Parallel Phase 2 Clinical Trial of Atezolizumab With or Without Low Dose Local Radiotherapy (2 x 2Gy) in Patients With Relapsed/Refractory Advanced Stage Follicular Lymphoma
Brief Title: Study of the PD-L1 Inhibitor Atezolizumab With or Without Low-dose, Local Radiation in Patients With Relapsed or Refractory Advanced Stage Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual and lack of funding.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-360
Record Dates: First submitted 2018-03-09; First posted 2018-03-14 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2019-12

CONDITIONS: Lymphoma
Keywords: Advanced Stage Follicular Lymphoma; Relapsed; Refractory; Atezolizumab; Dose Local Radiotherapy (2 x 2Gy); 17-360
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel, open-label, phase II clinical trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- atezolizumab (Experimental): All patients will receive open-label atezolizumab 1200mg IV on day 1 of a 21-day cycle for a planned total of 17 cycles of therapy (1 year).
  Interventions: Drug: atezolizumab
- atezolizumab plus low-dose, local radiotherapy (Experimental): All patients will receive open-label atezolizumab 1200mg IV on day 1 of a 21-day cycle for a planned total of 17 cycles of therapy (1 year). 4Gy will be administered in 2 fractions to a single nodal site amenable to radiation as identified by the radiation oncologist on day 2 and day 3 of Cycle 1 (over the two days following to the first dose of atezolizumab ).
  Interventions: Drug: atezolizumab; Radiation: Low- Dose, Local Radiotherapy

INTERVENTIONS:
Drug: atezolizumab — 1200mg IV on day 1 of a 21-day cycle for a planned total of 17 cycles of therapy (1 year).
Radiation: Low- Dose, Local Radiotherapy — 4Gy will be administered in 2 fractions to a single nodal site amenable to radiation as identified by the radiation oncologist on day 2 and day 3 of Cycle 1 (over the two days following to the first dose of atezolizumab ).
  Arms: atezolizumab plus low-dose, local radiotherapy

SUMMARY:
The purpose of this study is to compare the safety and effects of atezolizumab with low dose radiation on people with relapsed or refractory follicular lymphoma, In this study, the patient will get either atezolizumab with low dose radiation or, atezolizumab alone. To be better, the atezolizumab and low dose radiation should increase life by 1 year or more compared to the usual approach.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF) Ability and willingness to comply with the requirements of the study protocol
* Age ≥ 18 years
* Relapsed or refractory follicular lymphoma grade 1, 2, or 3A

  * Relapsed disease is defined as having relapsed after greater than 6 months of prior treatment for follicular lymphoma
  * Refractory disease is defined as failure to achieve a complete response or relapsed within 6 months of treatment for follicular lymphoma
  * Pretreatment biopsy for fresh tumor tissue collection is required
  * If patient has recently undergone a biopsy and has not received any intercurrent anti-lymphoma therapy, archival tissue can be used
* Stage III/IV disease

  ° Stage II disease is also eligible if disease is not encompassible within a single radiation field, as determined by the radiation oncologist
* At least 1 prior treatment for follicular lymphoma (no restriction to number or type of prior therapies)

  * Patient treated for transformed diffuse large B cell lymphoma (DLBCL) who have retrograde transformation are eligible provided they have received at least one prior treatment for the follicular lymphoma
* Site of disease amenable to low-dose, local radiotherapy (2 x 2Gy), as recommended by the radiation oncologist
* At least one bi-dimensionally measurable nodal lesion > 1.5 cm in its longest diameter by CT scan or magnetic resonance imaging, as defined by the Lugano Classification
* Adequate hematologic and end organ function:

  * ANC ≥ 1500 cells/µL
  * If there is documented bone marrow involvement of follicular lymphoma, ANC must be >/= 1000 cells/µL
  * Platelet count ≥ 75,000/µL
  * If there is documented bone marrow involvement of follicular lymphoma, platelet count must be >/= 50,000/µL
  * Hemoglobin ≥ 9.0 g/dL
  * If there is documented bone marrow involvement of follicular lymphoma, hemoglobin must be >/= 8.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
  * AST and ALT ≤ 3.0 x ULN
  * Patients with liver involvement: AST and/or ALT ≤ 5 x ULN Alkaline phosphatase ≤ 2.5 x ULN
  * Patients with documented liver involvement or bone metastases:

alkaline phosphatase ≤ 5 x ULN

* Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation:

  (140 - age) x (weight in kg) x (0.85 if female) 72 x (serum creatinine in mg/dL)
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use for 5 months after the last dose of ATEZOLIZUMAB. Women must refrain from donating eggs during this same period

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>/= 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Mullerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
  * Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. If required per local guidelines or regulations, locally recognized acceptable methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Willingness to undergo on-treatment biopsies unless not clinically feasible while on treatment

Exclusion Criteria:

* Follicular lymphoma grade 3B
* Concurrent aggressive non-Hodgkin lymphoma (e.g. diffuse large B cell lymphoma [DLBCL])
* Any anticancer therapy, including chemotherapy, hormonal therapy, investigational therapy, or radiotherapy, within 3 weeks, or 5 half lifes, whichever is shortest, prior to initiation of study treatment. However, the following are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy, provided it is discontinued at least 1 week prior to Cycle 1, Day 1
  * Palliative radiotherapy for bone metastases, provided most recent fraction not given within 2 weeks of Cycle 1, Day 1 and most recent fraction was not administered to planned area of radiation while on study.
* AEs from prior anticancer therapy that have not resolved to Grade ≤ 1 with exception of alopecia or skin/nail hyperpigmentation
* Bisphosphonate therapy for symptomatic hypercalcemia within 2 weeks of cycle 1, day 1

  ° Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed. Denosumab should not be used while on therapy
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Active central nervous system (CNS) involvement of lymphoma

  ° Patients with a history of CNS involvement of lymphoma are eligible, provided they received treatment greater than 30 days prior to cycle 1 day 1 and there is no evidence of involvement on most recent assessment
* Pregnant, or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment.

  ° Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment
* Known hypersensitivity to Chinese hamster ovary cell products, other recombinant human antibodies, or to any component of the atezolizumab formulation
* Inability to comply with study and follow-up procedures
* Active or history of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener"s granulomatosis, Sjögren"s syndrome, Bell"s palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
  * Patients with inactive inflammatory bowel disease, not currently receiving therapy, may be eligible.
  * Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
  * Rash must cover less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
  * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  °History of radiation pneumonitis is permitted provided patient is asymptomatic and did not require systemic or inhaled corticosteroids for treatment of symptomatic radiation pneumonitis
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active tuberculosis
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1, within 5 months after the final dose, or anticipation that such a live, attenuated vaccine will be required during the study

  ° Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* Malignancies other than the disease under study within 3 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate-specific antigen [PSA] ≤ 10 mg/mL, etc.)

Medication-Related Exclusion Criteria:

* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents. Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met:

  * Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose
  * No history of severe immune-related adverse effects from ant-CTLA-4 (NCI CTCAE Grade 3 and 4)
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]-a of interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
* Treatment with systemic immunosuppressive medication (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 1 week prior to Cycle 1, Day 1.

  * Patient who have received acute, low-dose systemic immunosuppressant medication (e.g., a one-time dose of dexamethasone for nausea or prednisone for intravenous contrast allergy) may be enrolled
  * Palliative systemic steroids for palliation of disease are allowed but must be discontinued at least 7 days prior to cycle 1, day 1
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Lia Palomba, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atezolizumab | Atezolizumab Plus Low-dose, Local Radiotherapy
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disease progression | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated early due to lack of funding and low accruals.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab | Atezolizumab Plus Low-dose, Local Radiotherapy | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 67 [67 to 67] | 39 [39 to 39] | 53 [39 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: objective response defined as CR or PR; as measured in non-irradiated sites of disease. Response will be assessed by the investigator per the Lugano Classification.
Time Frame: 3 years
Population: Data were not collected
Arm/Group | Atezolizumab | Atezolizumab Plus Low-dose, Local Radiotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: N/A - Data were not collected
Description: Study was terminated due to lack of funding and low accrual rate.
Arm/Group | Atezolizumab | Atezolizumab Plus Low-dose, Local Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03465891/Prot_SAP_000.pdf